CLINICAL TRIAL: NCT03446612
Title: A Randomized, Repeat Dose, Open Label, Parallel Group, Multi-center Study to Evaluate the Effect of Daprodustat Compared to Darbepoetin Alfa on Forearm Blood Flow in Participants With Anemia of Chronic Kidney Disease That Are Not Dialysis Dependent
Brief Title: Anemia Study in Chronic Kidney Disease (CKD) : Erythropoiesis Via a Novel Prolyl Hydroxylase Inhibitor (PHI) Daprodustat -Forearm Blood Flow (ASCEND-FBF)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study is terminated due to feasibility in recruitment.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 205767; 2017-002268-42 (EudraCT Number)
Record Dates: First submitted 2018-02-20; First posted 2018-02-27 (Actual); Results first posted 2021-07-21 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Anaemia
Keywords: darbepoetin alpha; challenge agents; daprodustat; FBF-CKD
MeSH Terms: conditions — Anemia | interventions — GSK1278863; Darbepoetin alfa; Acetylcholine; Nitroprusside; omega-N-Methylarginine

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either daprodustat or darbepoetin alfa. A central randomization approach will be used with stratification by center.
Masking Description: This is an open-label study. However, a central FBF reader, who will read and evaluate the FBF data, will be blinded to the treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants receiving Daprodustat (Experimental): Participants will receive 2 milligram (mg) daprodustat tablets once daily via oral route for a period of 41 days.
  Interventions: Drug: Daprodustat; Drug: Acetylcholine; Drug: Sodium nitroprusside; Drug: L-N-monomethyl arginine acetate (L-NMMA)
- Participants receiving Darbepoetin alfa (Active Comparator): Participants will receive Darbepoetin alfa solution for injection, administered as a single subcutaneous injection, once every two weeks (Days 1, 14 and 28).
  Interventions: Drug: Darbepoetin alfa; Drug: Acetylcholine; Drug: Sodium nitroprusside; Drug: L-N-monomethyl arginine acetate (L-NMMA)

INTERVENTIONS:
Drug: Daprodustat — Daprodustat will be available as 1 mg, 2 mg and 4 mg oral tablets. Daprodustat will be administered once daily by oral route without regard for food.
  Arms: Participants receiving Daprodustat
Drug: Darbepoetin alfa — Darbepoetin alfa will be given as solution for injection for subcutaneous administration every 2 weeks.
  Arms: Participants receiving Darbepoetin alfa
Drug: Acetylcholine — Acetylcholine will be used as a challenge agent and will be infused at 7.5, 15 and 30 micrograms/minute each for 6 minutes per infusion into the brachial artery of the test arm.
Drug: Sodium nitroprusside — Sodium nitroprusside will be used as a challenge agent and will be infused at 3 and 10 micrograms/minute each for 6 minutes per infusion into the brachial artery of the test arm.
Drug: L-N-monomethyl arginine acetate (L-NMMA) — L-N-monomethyl arginine acetate will be used as a challenge agent and will be infused at a doses of 2 and 8 micromoles/minute for 6 minutes into the brachial artery of the test arm.

SUMMARY:
Daprodustat has demonstrated an ability to effectively raise hemoglobin concentrations with lower erythropoietin (EPO) levels than those observed after administration of recombinant human erythropoietin (rhEPOs). Therefore, daprodustat has the potential to treat anemia of chronic kidney disease (CKD) with a lower cardiovascular (CV) risk than is observed with the rhEPOs. While the effect of rhEPOs on endothelial function has been assessed, to date the effect of daprodustat or other prolyl hydroxylase inhibitor (PHI) compounds on endothelial function has not. Therefore, the purpose of this study is to compare the effect of daprodustat to darbepoetin alfa on endothelial function by assessing FBF in participants with anemia of CKD by using venous occlusion plethysmography as a means to estimate the potential for daprodustat to have a lower risk of CV events as compared to rhEPO.

This study will use a randomized, repeat dose, open label, parallel group design, in adult, not on-dialysis, male and female participants with anemia of CKD that are currently not treated with rhEPOs.

The study will comprise of three study periods: a screening period starting up to 30 days prior to Day 1, a 42 day (6 week) treatment period, and a follow-up visit up to 14 days later. The total duration of participants involvement is up to 14 weeks (including screening and follow up visit). Approximately 50 participants will be randomized to either daprodustat or darbepoetin alfa.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be at least 18 years of age inclusive, at the time of signing the informed consent.
* Participants who are Stage 3, 4 or 5 CKD defined by estimated Glomerular Filtration Rate (eGFR) using the CKD Epidemiology Collaboration (CKD-EPI) formula.
* Hemoglobin as measured by HemoCue at screening visit and Day 1 is <=11.0 grams/deciliter (g/dL) [<=110 gram/Litre (g/L)].
* Palpable brachial artery as assessed at screening.
* Participants, if necessary may be on stable maintenance oral iron supplementation (<50% change in overall dose and compliance of 80% of prescribed doses in the 4 weeks prior to and including the screening period). If participants have been on intravenous (IV) iron, then participants will not have received IV iron for 4 weeks prior to the Day 1 visit.
* Male or female participants will be included.
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: Not a woman of childbearing potential (WOCBP) or a WOCBP who has been on an approved form of contraceptive for the 4 weeks prior to Day 1 and agrees to follow the contraceptive guidance until the Follow-up visit.
* Capable of giving signed informed consent.

Exclusion Criteria:

* On dialysis or clinical evidence of impending need to initiate dialysis within 12 weeks of Day 1.
* Planned kidney transplant within 12 weeks of Day 1.
* Presence of an arteriovenous (AV) fistula.
* Recombinant human erythropoietin use within the 12 weeks prior to the screening visit and through Day 1.
* History of severe allergic or anaphylactic reactions or hypersensitivity to the study treatment or challenge agents, or excipients in the study treatments or challenge agents.
* Planned use of any prescription or non-prescription drugs or dietary supplements that are prohibited from screening until all assessments on Day 42 have been successfully completed.
* The participant has participated in a clinical trial and has received an experimental investigational product within the prior 30 days or within 5 half-lives of the investigational product (whichever is longer) prior to screening and through Day 1.
* At or below the lower limit of the reference range at screening for Vitamin B12 (may rescreen in a minimum of 8 weeks).
* Ferritin <=50 nanograms/milliliter [<=50 microgram/liter (µg/L)] at screening.
* Transferrin saturation (TSAT) <=15% (0.15) at screening.
* Folate <2.0 nanogram/milliliter (4.5 nanomoles/liter; may rescreen in a minimum of 8 weeks) at screening.
* High sensitivity C-reactive protein (hs-CRP) >=50 micrograms/milliliter (>=50 mg/L) at screening.
* Myocardial infarction or acute coronary syndrome <=12 weeks prior to screening and through Day 1.
* Hospitalization for greater than 24 hours <=12 weeks prior to screening and through Day 1.
* Stroke or transient ischemic attack <=12 weeks prior to screening and through Day 1.
* Class 4 heart failure, as defined by the New York Heart Association (NYHA) functional classification system.
* Resting SBP >180 millimeters of mercury (mmHg) or DBP >110 mmHg at screening visit or current uncontrolled hypertension as determined by the investigator.
* QT interval corrected for heart rate using Bazett's formula (QTcB) >500 milliseconds (msec), or QTcB >530 msec in participants with bundle branch block. There is no corrected QT (QTc) exclusion for participants with a predominantly ventricular paced rhythm.
* Active chronic inflammatory disease that could impact erythropoiesis.
* History of bone marrow aplasia or pure red cell aplasia.
* Conditions, other than anemia of CKD, which can affect erythropoiesis.
* Evidence of actively bleeding gastric, duodenal, or esophageal ulcer disease or clinically significant gastrointestinal bleeding from <=8 weeks prior to screening and through Day 1.
* ALT >2 times upper limit of normal (ULN; screening only).
* Bilirubin >1.5 times ULN (screening only); Isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Major surgery within the 12 weeks prior to screening and through Day 1, or planned during the study.
* Anticipated or planned vascular access surgery (i.e., arteriovenous [AV] fistula) within the 12 weeks prior to screening and through the Day 42 assessments.
* Received a tissue heart valve replacement or repair within the 6 months prior to screening or has received a mechanical heart valve replacement.
* Blood transfusion within 6 weeks prior to screening and through Day 1, or an anticipated need for blood transfusion during the study.
* Clinical evidence of an acute infection, or history of infection requiring IV antibiotic therapy from 8 weeks prior to screening and through Day 1. Prophylactic oral antibiotics are allowed.
* History of malignancy within the two years prior to screening and through Day 1 or currently receiving treatment for cancer, with the exception of localized squamous cell or basal cell carcinoma of the skin definitively treated 12 weeks prior to Day 1.
* Platelet count <50,000/µL (<50 Giga cells per liter).
* History of a bleeding disorder (e.g., hemophilia).
* Any other condition, clinical or laboratory abnormality, or examination finding that the investigator considers would put the participant at unacceptable risk, which may affect study compliance or prevent understanding of the aims or investigational procedures or possible consequences of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-05-29 (Actual); Study Completion 2019-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United Kingdom (3):
  - GSK Investigational Site, Cambridge, Cambridgeshire
  - GSK Investigational Site, Edinburgh
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open label, parallel group study that evaluated the effect of daprodustat and darbepoetin alfa on forearm blood flow (FBF) in participants with anemia of chronic kidney disease that are not dialysis dependent.
Pre-assignment Details: Participants were enrolled in multiple centers in United Kingdom. A total of 6 participants were enrolled in the study and only 5 participants were randomized to receive study treatment.
Groups:
- Daprodustat: Participants were randomized to receive 2 milligram (mg) daprodustat tablets once daily via oral route for a period of 41 days.
- Darbepoetin Alfa: Participants were randomized to receive darbepoetin alfa solution for injection, administered as a single subcutaneous injection, once every two weeks (Days 1, 14 and 28).
Period: Overall Study
Arm/Group | Daprodustat | Darbepoetin Alfa
Started | 2 | 3
Completed | 2 | 2
Not Completed | 0 | 1
Not completed — Protocol defined stopping criteria | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Daprodustat | Darbepoetin Alfa | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.0 (2.83) | 53.0 (15.72) | 56.6 (12.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian/European Heritage | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in FBF Ratio in Response to Acetylcholine (Day 1 to Day 42)
Description: Venous occlusion plethysmography was used for FBF assessment. Acetylcholine (ACH) was infused intra-arterially at 7.5, 15 and 30 micrograms/minute (ug/min) each for 6 minutes per infusion. FBF ratio was defined as the ratio of a participant's treatment (infused) arm value divided by the non-treatment (non-infused) arm value. The overall ratio was determined by taking the participant's Day 42 FBF ratio and dividing by the Day 1 FBF ratio.
Time Frame: Day 1 to Day 42
Population: Pharmacodynamic Per-Protocol (PDPP) population included all randomized participants who provided pharmacodynamic (PD) data at Day 1 and Day 42. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 2 | 2
Ratio
  ACH 7.5 ug/min, n=2, 2 | 1.1304 (0.30030) | 0.4351 (0.17032)
  ACH 15 ug/min, n=1, 2: number analyzed (Participants) | 1 | 2
  ACH 15 ug/min, n=1, 2 | 0.7866 (NA) — Not applicable (NA) indicates standard deviation could not be calculated as a single participant was analyzed. | 0.6183 (0.00435)
  ACH 30 ug/min, n=1, 2: number analyzed (Participants) | 1 | 2
  ACH 30 ug/min, n=1, 2 | 1.1328 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | 0.8090 (0.28395)
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Other; FBF ratio difference = 0.6953, Standard Deviation 0.12998 — The difference between daprodustat and darbepoetin alfa FBF ratio in response to acetylcholine (7.5 ug/min) is presented
Statistical Analysis 2: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Other; FBF ratio difference = 0.1683 — The difference between daprodustat and darbepoetin alfa FBF ratio in response to acetylcholine (15 ug/min) is presented
Statistical Analysis 3: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Other; FBF ratio difference = 0.3238 — The difference between daprodustat and darbepoetin alfa FBF ratio in response to acetylcholine (30 ug/min) is presented

2. Secondary Outcome: Change in the Absolute FBF From Day 1 to Day 42 in Response to Acetylcholine
Description: Venous occlusion plethysmography was used for FBF assessment. Acetylcholine was infused intra-arterially at 7.5, 15 and 30 ug/min each for 6 minutes per infusion. Measures were made in both arms concurrently. Change in the absolute FBF from Day 1 to Day 42 in response to acetylcholine is the difference between absolute value of FBF in infused arm on Day 1 and Day 42 in response to acetylcholine.
Time Frame: Day 1 to Day 42
Population: PDPP Population. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: ug/min
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 2 | 2
ug/min
  7.5 ug/min, n=2, 2 | 8.3180 (4.50592) | -6.0360 (3.09976)
  15 ug/min, n=1, 2: number analyzed (Participants) | 1 | 2
  15 ug/min, n=1, 2 | -4.6374 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | -8.8299 (9.98143)
  30 ug/min, n=1, 2: number analyzed (Participants) | 1 | 2
  30 ug/min, n=1, 2 | -2.6735 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | -4.5121 (5.66731)

3. Secondary Outcome: Change in FBF Ratio in Response to Sodium Nitroprusside (Day 1 to Day 42)
Description: Venous occlusion plethysmography was used for FBF assessment. Sodium nitroprusside was infused at 3 and 10 ug/min each for 6 minutes per infusion into the brachial artery of the test arm. FBF ratio was defined as the ratio of a participant's treatment (infused) arm value divided by the non-treatment (non-infused) arm value. The overall ratio was determined by taking the participant's Day 42 FBF ratio and dividing by the Day 1 FBF ratio.
Time Frame: Day 1 to Day 42
Population: PDPP Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1 | 2
Ratio
  3 ug/min | 1.0388 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | 0.7420 (0.07407)
  10 ug/min | 2.1447 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | 0.7022 (0.00860)
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Other; FBF ratio difference = 0.2968 — The difference between daprodustat and darbepoetin alfa FBF ratio in response to sodium nitroprusside (3 ug/min) is presented
Statistical Analysis 2: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Other; FBF ratio difference = 1.4425 — The difference between daprodustat and darbepoetin alfa FBF ratio in response to sodium nitroprusside (10 ug/min) is presented

4. Secondary Outcome: Change in the Absolute FBF From Day 1 to Day 42 in Response to Sodium Nitroprusside
Description: Venous occlusion plethysmography was used for FBF assessment. Sodium nitroprusside was infused at 3 and 10 ug/min each for 6 minutes per infusion into the brachial artery of the test arm. Measures were made in both arms concurrently. Change in the absolute FBF from Day 1 to Day 42 in response to sodium nitroprusside is the difference between absolute value of FBF in infused arm on Day 1 and Day 42 in response to sodium nitroprusside.
Time Frame: Day 1 to Day 42
Population: PDPP Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: ug/min
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1 | 2
ug/min
  3 ug/min | -0.2560 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | 0.3844 (0.52197)
  10 ug/min | 6.8103 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | -0.2873 (1.11519)

5. Secondary Outcome: Change in FBF Ratio in Response to NG-monomethyl Arginine Acetate (L-NMMA) (Day 1 to Day 42)
Description: Venous occlusion plethysmography was used for FBF assessment. Effects on basal nitric oxide synthesis was assessed using L-NMMA at doses of 2 and 8 micromoles per minute (umol/min) each infused for 6 minutes into the brachial artery of the test arm. FBF ratio was defined as the ratio of a participant's treatment (infused) arm value divided by the non-treatment (non-infused) arm value. The overall ratio was determined by taking the participant's Day 42 FBF ratio and dividing by the Day 1 FBF ratio.
Time Frame: Day 1 to Day 42
Population: PDPP Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1 | 1
Ratio
  2 umol/min | 0.7426 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | 0.9024 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
  8 umol/min | 0.4975 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | 0.8690 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Other; FBF ratio difference = -0.1598 — The difference between daprodustat and darbepoetin alfa FBF ratio in response to L-NMMA (2 umol/min) is presented
Statistical Analysis 2: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Other; FBF ratio difference = -0.3715 — The difference between daprodustat and darbepoetin alfa FBF ratio in response to L-NMMA (8 umol/min) is presented

6. Secondary Outcome: Change in the Absolute FBF From Day 1 to Day 42 in Response to L-NMMA
Description: Venous occlusion plethysmography was used for FBF assessment. Effects on basal nitric oxide synthesis was assessed using L-NMMA at doses of 2 and 8 umol/min each infused for 6 minutes into the brachial artery of the test arm. Measures were made in both arms concurrently. Change in the absolute FBF from Day 1 to Day 42 in response to L-NMMA is the difference between absolute value of FBF in infused arm on Day 1 and Day 42 in response to L-NMMA.
Time Frame: Day 1 to Day 42
Population: PDPP Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: umol/min
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1 | 1
umol/min
  2 umol/min | 1.1508 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | 0.3558 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
  8 umol/min | 0.0974 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | 0.0399 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.

7. Secondary Outcome: Change in FBF Ratio in Response to Acetylcholine at Day 42 Versus (vs) Day 1 in Participants Treated With Daprodustat
Description: Venous occlusion plethysmography was used for FBF assessment. Acetylcholine was infused intra-arterially at 7.5, 15 and 30 ug/min each for 6 minutes per infusion. The Day 42 ratio was calculated by taking the participants Day 42 treatment (infused) arm and dividing by the Day 42 non-treatment (control) arm value. The Day 1 ratio was calculated by taking the participants Day 1 treatment (infused) arm and dividing by the Day 1 non-treatment (control) arm value. Change in FBF ratio from Day 1 to Day 42 was determined by taking the participants Day 42 ratio and dividing by the Day 1 ratio.
Time Frame: Day 1 and Day 42
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Daprodustat
Number analyzed (Participants) | 2
Ratio
  7.5 ug/min, n=2 | 0.2744 (0.91996)
  15 ug/min, n=1: number analyzed (Participants) | 1
  15 ug/min, n=1 | -0.8503 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed
  30 ug/min, n=1: number analyzed (Participants) | 1
  30 ug/min, n=1 | 0.5482 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed

8. Secondary Outcome: Change in FBF Ratio in Response to Sodium Nitroprusside at Day 42 vs Day 1 in Participants Treated With Daprodustat
Description: Venous occlusion plethysmography was used for FBF assessment. Sodium nitroprusside was infused at 3 and 10 ug/min each for 6 minutes per infusion into the brachial artery of the test arm. The Day 42 ratio was calculated by taking the participants Day 42 treatment (infused) arm and dividing by the Day 42 non-treatment (control) arm value. The Day 1 ratio was calculated by taking the participants Day 1 treatment (infused) arm and dividing by the Day 1 non-treatment (control) arm value. Change in FBF ratio from Day 1 to Day 42 was determined by taking the participants Day 42 ratio and dividing by the Day 1 ratio.
Time Frame: Day 1 and Day 42
Population: PDPP Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Daprodustat
Number analyzed (Participants) | 1
Ratio
  3 ug/min | 0.1618 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
  10 ug/min | 3.2651 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.

9. Secondary Outcome: Change in FBF Ratio in Response to L-NMMA at Day 42 vs Day 1 in Participants Treated With Daprodustat
Description: Venous occlusion plethysmography was used for FBF assessment. Effects on basal nitric oxide synthesis was assessed using L-NMMA at doses of 2 and 8 umol/min each infused for 6 minutes into the brachial artery of the test arm. The Day 42 ratio was calculated by taking the participants Day 42 treatment (infused) arm and dividing by the Day 42 non-treatment (control) arm value. The Day 1 ratio was calculated by taking the participants Day 1 treatment (infused) arm and dividing by the Day 1 non-treatment (control) arm value. Change in FBF ratio from Day 1 to Day 42 was determined by taking the participants Day 42 ratio and dividing by the Day 1 ratio.
Time Frame: Day 1 and Day 42
Population: PDPP Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Daprodustat
Number analyzed (Participants) | 1
Ratio
  2 umol/min | -0.3896 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
  8 umol/min | -0.7216 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.

10. Secondary Outcome: Change in FBF Ratio in Response to Acetylcholine at Day 42 vs Day 1 in Participants Treated With Darbepoetin Alfa
Description: as for outcome 7
Time Frame: Day 1 and Day 42
Population: PDPP Population
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Darbepoetin Alfa
Number analyzed (Participants) | 2
Ratio
  7.5 ug/min | -2.0376 (0.63291)
  15 ug/min | -1.4559 (0.01558)
  30 ug/min | -1.0652 (1.56389)

11. Secondary Outcome: Change in FBF Ratio in Response to Sodium Nitroprusside at Day 42 vs Day 1 in Participants Treated With Darbepoetin Alfa
Description: as for outcome 8
Time Frame: Day 1 and Day 42
Population: PDPP Population.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Darbepoetin Alfa
Number analyzed (Participants) | 2
Ratio
  3 ug/min | -0.7503 (0.26692)
  10 ug/min | -1.2405 (0.15366)

12. Secondary Outcome: Change in FBF Ratio in Response to L-NMMA at Day 42 vs Day 1 in Participants Treated With Darbepoetin Alfa
Description: as for outcome 9
Time Frame: Day 1 and Day 42
Population: PDPP Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Darbepoetin Alfa
Number analyzed (Participants) | 1
Ratio
  2 umol/min | -0.081 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
  8 umol/min | -0.1351 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.

13. Secondary Outcome: Change in the Absolute FBF in Response to Acetylcholine at Day 42 vs Day 1 in Participants Treated With Daprodustat
Description: Venous occlusion plethysmography was used for FBF assessment. Acetylcholine was infused intra-arterially at 7.5, 15 and 30 ug/min each for 6 minutes per infusion. Measures were made in both arms concurrently. Change in the absolute FBF in response to acetylcholine at Day 42 vs Day1 is the difference between absolute value of FBF in infused arm on Day 1 and Day 42 in response to acetylcholine in participants treated with daprodustat.
Time Frame: Day 1 and Day 42
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ug/min
Arm/Group | Daprodustat
Number analyzed (Participants) | 2
ug/min
  7.5 ug/min, n=2 | 8.3180 (4.50592)
  15 ug/min, n=1: number analyzed (Participants) | 1
  15 ug/min, n=1 | -4.6374 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
  30 ug/min, n=1: number analyzed (Participants) | 1
  30 ug/min, n=1 | -2.6735 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.

14. Secondary Outcome: Change in the Absolute FBF in Response to Sodium Nitroprusside at Day 42 vs Day 1 in Participants Treated With Daprodustat
Description: Venous occlusion plethysmography was used for FBF assessment. Sodium nitroprusside was infused at 3 and 10 ug/min each for 6 minutes per infusion into the brachial artery of the test arm. Measures were made in both arms concurrently. Change in the absolute FBF in response to sodium nitroprusside at Day 42 vs Day 1 is the difference between absolute value of FBF in infused arm on Day 1 and Day 42 in response to sodium nitroprusside in participants treated with daprodustat.
Time Frame: Day 1 and Day 42
Population: PDPP Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: ug/min
Arm/Group | Daprodustat
Number analyzed (Participants) | 1
ug/min
  3 ug/min | -0.2560 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
  10 ug/min | 6.8103 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.

15. Secondary Outcome: Change in the Absolute FBF in Response to L-NMMA at Day 42 vs Day 1 in Participants Treated With Daprodustat
Description: Venous occlusion plethysmography was used for FBF assessment. Effects on basal nitric oxide synthesis was assessed using L-NMMA at doses of 2 and 8 umol/min each infused for 6 minutes into the brachial artery of the test arm. Measures were made in both arms concurrently. Change in the absolute FBF in response to L-NMMA at Day 42 vs Day 1 is the difference between absolute value of FBF in infused arm on Day 1 and Day 42 in response to L-NMMA in participants treated with daprodustat.
Time Frame: Day 1 and Day 42
Population: PDPP Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: umol/min
Arm/Group | Daprodustat
Number analyzed (Participants) | 1
umol/min
  2 umol/min | 1.1508 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
  8 umol/min | 0.0974 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.

16. Secondary Outcome: Change in the Absolute FBF in Response to Acetylcholine at Day 42 vs Day 1 in Participants Treated With Darbepoetin Alfa
Description: Venous occlusion plethysmography was used for FBF assessment. Acetylcholine was infused intra-arterially at 7.5, 15 and 30 ug/min each for 6 minutes per infusion. Measures were made in both arms concurrently. Change in the absolute FBF in response to acetylcholine at Day 42 vs Day1 is the difference between absolute value of FBF in infused arm on Day 1 and Day 42 in response to acetylcholine in participants treated with darbepoetin alfa.
Time Frame: Day 1 and Day 42
Population: PDPP Population
Measure: Mean (Standard Deviation); unit: ug/min
Arm/Group | Darbepoetin Alfa
Number analyzed (Participants) | 2
ug/min
  7.5 ug/min | -6.0360 (3.09976)
  15 ug/min | -8.8299 (9.98143)
  30 ug/min | -4.5121 (5.66731)

17. Secondary Outcome: Change in the Absolute FBF in Response to Sodium Nitroprusside at Day 42 vs Day 1 in Participants Treated With Darbepoetin Alfa
Description: Venous occlusion plethysmography was used for FBF assessment. Sodium nitroprusside was infused at 3 and 10 ug/min each for 6 minutes per infusion into the brachial artery of the test arm. Measures were made in both arms concurrently. Change in the absolute FBF in response to sodium nitroprusside at Day 42 vs Day 1 is the difference between absolute value of FBF in infused arm on Day 1 and Day 42 in response to sodium nitroprusside in participants treated with darbepoetin alfa.
Time Frame: Day 1 and Day 42
Population: PDPP Population
Measure: Mean (Standard Deviation); unit: ug/min
Arm/Group | Darbepoetin Alfa
Number analyzed (Participants) | 2
ug/min
  3 ug/min | 0.3844 (0.52197)
  10 ug/min | -0.2873 (1.11519)

18. Secondary Outcome: Change in the Absolute FBF in Response to L-NMMA at Day 42 vs Day 1 in Participants Treated With Darbepoetin Alfa
Description: Venous occlusion plethysmography was used for FBF assessment. Effects on basal nitric oxide synthesis was assessed using L-NMMA at doses of 2 and 8 umol/min each infused for 6 minutes into the brachial artery of the test arm. Measures were made in both arms concurrently. Change in the absolute FBF in response to L-NMMA at Day 42 vs Day 1 is the difference between absolute value of FBF in infused arm on Day 1 and Day 42 in response to L-NMMA in participants treated with darbepoetin alfa.
Time Frame: Day 1 and Day 42
Population: PDPP Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: umol/min
Arm/Group | Darbepoetin Alfa
Number analyzed (Participants) | 1
umol/min
  2 umol/min | 0.3558 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
  8 umol/min | 0.0399 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.

19. Secondary Outcome: Change in Augmentation Index (AIx) From Day 1 to 42
Description: Pulse wave analysis (PWA) is a reproducible, noninvasive method for assessing AIx (a measure of the contribution that wave reflection makes to the arterial pressure waveform). The amplitude and timing of the reflected wave ultimately depends on the stiffness of the small (pre-resistance) vessels and large arteries, and thus, AIx provides a measure of systemic arterial stiffness. A high-fidelity micro manometer was used to obtain accurate readings of the peripheral pressure waveforms by flattening, but not occluding, the radial artery of the dominant arm using gentle pressure. AIx was defined as the augmentation (difference between systolic peaks) expressed as a percentage of the overall pulse pressure. Data for change in AIx from Day 1 to 42 was presented.
Time Frame: Day 1 to Day 42
Population: PDPP Population
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 2 | 2
Percentage | -3.000 (0.0000) | -4.000 (2.8284)

20. Secondary Outcome: Change in Pulse Wave Velocity (PWV) From Day 1 to Day 42
Description: PWV was assessed with a high-fidelity micro manometer which was used to obtain accurate readings of the peripheral pressure waveforms by flattening, but not occluding, the carotid and femoral arteries as the two points of measure. Data for change in PWV from Day 1 to 42 was presented.
Time Frame: Day 1 to Day 42
Population: PDPP Population
Measure: Mean (Standard Deviation); unit: meters per second (m/sec)
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 2 | 2
meters per second (m/sec) | 2.075 (1.4496) | 0.100 (0.2828)

21. Secondary Outcome: Number of Participants With Any Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participants, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability, is a congenital anomaly/birth effect.
Time Frame: Up to 59 days
Population: Safety Population includes all randomised participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 2 | 3
Participants
  Any AEs | 0 | 1
  Any SAEs | 0 | 0

22. Secondary Outcome: Number of Participants With Any AE of Special Interest (AESI)
Description: AESIs were identified based on non-clinical studies with daprodustat, clinical experience with recombinant human erythropoietins (rhEPOs), and current information regarding hypoxia-inducible factor (HIF)-regulated pathways in mediating hypoxia-associated pathophysiology. The AESIs for daprodustat were identified as follows: Thrombosis and/or tissue ischemia secondary to excessive erythropoiesis; Death, MI, stroke, heart failure, thromboembolic events, thrombosis of vascular access; Cardiomyopathy; Pulmonary artery hypertension; Cancer-related mortality and tumor progression and recurrence Esophageal and gastric erosions; Proliferative retinopathy, macular edema, choroidal neovascularization; Exacerbation of rheumatoid arthritis and Worsening of hypertension.
Time Frame: Up to 59 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 2 | 3
Participants | 0 | 0

23. Secondary Outcome: Number of Participants Discontinuing the Randomized Study Treatment
Description: Number of participants who discontinued the randomized study treatment were assessed.
Time Frame: Up to Day 42
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 2 | 3
Participants | 0 | 0

24. Other Pre Specified Outcome: Absolute Values of Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP)
Description: DBP and SBP were measured in a semi-supine position with a completely automated device preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions.
Time Frame: Days 1, 14, 28, 42 and 59
Population: Safety Population. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 2 | 3
millimeters of mercury (mmHg)
  DBP, Day 1, n=2, 3 | 73.5 (13.44) | 69.3 (13.05)
  DBP, Day 14, n=2, 3 | 67.0 (5.66) | 74.3 (13.05)
  DBP, Day 28, n=2, 3 | 73.5 (7.78) | 79.3 (25.54)
  DBP, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  DBP, Day 42, n=2, 2 | 76.0 (9.90) | 73.0 (8.49)
  DBP, Day 59, n=2, 3 | 69.5 (9.19) | 82.7 (18.15)
  SBP, Day 1, n=2, 3 | 144.0 (43.84) | 134.3 (18.34)
  SBP, Day 14, n=2, 3 | 130.0 (28.28) | 127.7 (23.25)
  SBP, Day 28, n=2, 3 | 135.5 (12.02) | 147.3 (39.63)
  SBP, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  SBP, Day 42, n=2, 2 | 145.5 (33.23) | 148.0 (45.25)
  SBP, Day 59, n=2, 3 | 135.5 (31.82) | 142.3 (29.14)

25. Other Pre Specified Outcome: Change From Baseline in DBP and SBP
Description: DBP and SBP were measured in a semi-supine position with a completely automated device preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline value (Day 1) is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and at Days 14, 28, 42 and 59
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 2 | 3
mmHg
  DBP, Day 14, n=2, 3 | -6.5 (7.78) | 5.0 (0.00)
  DBP, Day 28, n=2, 3 | 0.0 (21.21) | 10.0 (13.00)
  DBP, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  DBP, Day 42, n=2, 2 | 2.5 (3.54) | 10.5 (0.71)
  DBP, Day 59, n=2, 3 | -4.0 (4.24) | 13.3 (5.13)
  SBP, Day 14, n=2, 3 | -14.0 (15.56) | -6.7 (4.93)
  SBP, Day 28, n=2, 3 | -8.5 (31.82) | 13.0 (38.43)
  SBP, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  SBP, Day 42, n=2, 2 | 1.5 (10.61) | 10.5 (20.51)
  SBP, Day 59, n=2, 3 | -8.5 (12.02) | 8.0 (24.02)

26. Other Pre Specified Outcome: Absolute Values of Electrocardiogram (ECG) Mean Heart Rate
Description: Full 12-lead ECG were recorded with the participant in a semi-supine position to measure heart rate.
Time Frame: Days 1, 42 and 59
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 2 | 3
Beats per minute
  Day 1, n=2, 3 | 69.0 (2.83) | 70.0 (14.11)
  Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Day 42, n=2, 2 | 61.0 (14.14) | 62.0 (9.90)
  Day 59, n=2, 3 | 71.5 (9.19) | 73.7 (20.03)

27. Other Pre Specified Outcome: Change From Baseline in ECG Mean Heart Rate
Description: Full 12-lead ECG were recorded with the participant in a semi-supine position to measure heart rate. Baseline value (Day 1) is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and at Days 42 and 59
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 2 | 3
Beats per minute
  Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Day 42, n=2, 2 | -8.0 (11.31) | -0.5 (2.12)
  Day 59, n=2, 3 | 2.5 (12.02) | 3.7 (9.50)

28. Other Pre Specified Outcome: Absolute Values of ECG Parameters- PR Interval, QRS Interval, and QT Interval and QT Interval Corrected for Heart Rate Using Bazett's Formula (QTcB)
Description: Full 12-lead ECGs were recorded with the participant in a semi-supine position to measure PR interval, QRS duration, QT interval and QTcB, calculated (machine read or manually).
Time Frame: Days 1, 42 and 59
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 2 | 3
Milliseconds
  PR Interval, Day 1, n=2, 3 | 139.0 (1.41) | 181.7 (23.16)
  PR Interval, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  PR Interval, Day 42, n=2, 2 | 146.5 (7.78) | 192.5 (10.61)
  PR Interval, Day 59, n=2, 3 | 146.5 (2.12) | 182.0 (18.00)
  QRS Duration, Day 1, n=2, 3 | 87.0 (7.07) | 94.7 (5.03)
  QRS Duration, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  QRS Duration, Day 42, n=2, 2 | 88.5 (9.19) | 96.5 (10.61)
  QRS Duration, Day 59, n=2, 3 | 87.0 (9.90) | 95.3 (7.02)
  QT Interval, Day 1, n=2, 3 | 395.5 (6.36) | 391.3 (14.47)
  QT Interval, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  QT Interval, Day 42, n=2, 2 | 413.5 (20.51) | 388.0 (11.31)
  QT Interval, Day 59, n=2, 3 | 383.5 (44.55) | 382.3 (33.71)
  QTcB Interval, Day 1, n=2, 3 | 424.0 (1.41) | 420.7 (31.79)
  QTcB Interval, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  QTcB Interval, Day 42, n=2, 2 | 414.5 (27.58) | 393.0 (19.80)
  QTcB Interval, Day 59, n=2, 3 | 416.5 (21.92) | 417.3 (33.32)

29. Other Pre Specified Outcome: Change From Baseline in ECG Parameters- PR Interval, QRS Duration, and QT Interval and QTcB
Description: Full 12-lead ECGs were recorded with the participant in a semi-supine position to measure PR interval, QRS duration, QT (uncorrected) interval and QTcB, calculated (machine read or manually). Baseline value (Day 1) is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and at Days 42 and 59
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 2 | 3
Milliseconds
  PR Interval, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  PR Interval, Day 42, n=2, 2 | 7.5 (6.36) | -2.0 (19.80)
  PR Interval, Day 59, n=2, 3 | 7.5 (0.71) | 0.3 (16.86)
  QRS Duration, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  QRS Duration, Day 42, n=2, 2 | 1.5 (2.12) | 1.5 (3.54)
  QRS Duration, Day 59, n=2, 3 | 0.0 (2.83) | 0.7 (2.31)
  QT Interval, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  QT Interval, Day 42, n=2, 2 | 18.0 (14.14) | -7.0 (7.07)
  QT Interval, Day 59, n=2, 3 | -12.0 (50.91) | -9.0 (19.67)
  QTcB Interval, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  QTcB Interval, Day 42, n=2, 2 | -9.5 (26.16) | -9.5 (13.44)
  QTcB Interval, Day 59, n=2, 3 | -7.5 (20.51) | -3.3 (8.02)

30. Other Pre Specified Outcome: Absolute Values of the Hematology Parameters of Platelet Count, White Blood Cell (WBC) Count (Absolute), Basophils, Eosinophils, Lymphocytes, Monocytes and Neutrophils
Description: Blood samples were collected for the analysis of hematology parameters including platelet count, leukocytes, basophils, eosinophils, lymphocytes, monocytes and neutrophils.
Time Frame: Days 1, 42 and 59
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Giga cells per Liter
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 2 | 3
Giga cells per Liter
  Platelet count, Day 1, n=2, 3 | 199.0 (63.64) | 191.7 (68.13)
  Platelet count, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Platelet count, Day 42, n=2, 2 | 203.5 (57.28) | 121.5 (13.44)
  Platelet count, Day 59, n=2, 3 | 193.0 (41.01) | 50.08 (50.08)
  Leukocytes, Day 1, n=2, 3 | 5.05 (1.202) | 6.30 (2.117)
  Leukocytes, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Leukocytes, Day 42, n=2, 2 | 6.05 (2.616) | 5.75 (2.051)
  Leukocytes, Day 59, n=2, 3 | 5.30 (1.414) | 7.20 (2.261)
  Basophils, Day 1, n=2, 3 | 0.045 (0.0212) | 0.057 (0.0503)
  Basophils, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Basophils, Day 42, n=2, 2 | 0.045 (0.0212) | 0.045 (0.0212)
  Basophils, Day 59, n=2, 3 | 0.035 (0.0071) | 0.050 (0.0400)
  Eosinophils, Day 1, n=2, 3 | 0.295 (0.1485) | 0.230 (0.1353)
  Eosinophils, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Eosinophils, Day 42, n=2, 2 | 0.300 (0.1980) | 0.175 (0.0778)
  Eosinophils, Day 59, n=2, 3 | 0.245 (0.1485) | 0.220 (0.1311)
  Lymphocytes, Day 1, n=2, 3 | 1.160 (0.2404) | 2.037 (1.4989)
  Lymphocytes, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Lymphocytes, Day 42, n=2, 2 | 1.275 (0.2616) | 1.150 (0.4808)
  Lymphocytes, Day 59, n=2, 3 | 0.785 (0.3748) | 2.033 (1.3580)
  Monocytes, Day 1, n=2, 3 | 0.400 (0.0566) | 0.607 (0.3147)
  Monocytes, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Monocytes, Day 42, n=2, 2 | 0.415 (0.0071) | 0.445 (0.2192)
  Monocytes, Day 59, n=2, 3 | 0.415 (0.0778) | 0.563 (0.2574)
  Neutrophils, Day 1, n=2, 3 | 3.160 (1.3576) | 3.387 (0.2053)
  Neutrophils, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Neutrophils, Day 42, n=2, 2 | 4.010 (2.6870) | 3.970 (2.1920)
  Neutrophils, Day 59, n=2, 3 | 3.825 (1.0112) | 4.343 (1.0060)

31. Other Pre Specified Outcome: Change From Baseline in Hematology Parameters of Platelet Count, Leukocytes, Basophils, Eosinophils, Lymphocytes, Monocytes and Neutrophils
Description: Blood samples were collected for the analysis of hematology parameters including platelet count, WBC count (Absolute), basophils, eosinophils, lymphocytes, monocytes and neutrophils. Baseline value (Day 1) is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and at Days 42 and 59
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Giga cells per Liter
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 2 | 3
Giga cells per Liter
  Platelet count, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Platelet count, Day 42, n=2, 2 | 4.5 (6.36) | -51.0 (70.71)
  Platelet count, Day 59, n=2, 3 | -6.0 (22.63) | -26.3 (51.98)
  Leukocytes, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Leukocytes, Day 42, n=2, 2 | 1.00 (1.414) | 0.65 (2.616)
  Leukocytes, Day 59, n=2, 3 | 0.25 (0.212) | 0.90 (1.054)
  Basophils, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Basophils, Day 42, n=2, 2 | 0.000 (0.0000) | 0.015 (0.0071)
  Basophils, Day 59, n=2, 3 | -0.010 (0.0283) | -0.007 (0.0115)
  Eosinophils, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Eosinophils, Day 42, n=2, 2 | 0.005 (0.0495) | 0.015 (0.0071)
  Eosinophils, Day 59, n=2, 3 | -0.050 (0.0000) | -0.010 (0.0100)
  Lymphocytes, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Lymphocytes, Day 42, n=2, 2 | 0.115 (0.0212) | -0.040 (0.0424)
  Lymphocytes, Day 59, n=2, 3 | -0.375 (0.6152) | -0.003 (0.1443)
  Monocytes, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Monocytes, Day 42, n=2, 2 | 0.015 (0.0636) | 0.020 (0.2263)
  Monocytes, Day 59, n=2, 3 | 0.015 (0.0212) | -0.043 (0.0586)
  Neutrophils, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Neutrophils, Day 42, n=2, 2 | 0.850 (1.3294) | 0.670 (2.3900)
  Neutrophils, Day 59, n=2, 3 | 0.665 (0.3465) | 0.957 (1.0929)

32. Other Pre Specified Outcome: Absolute Values of the Hematology Parameter of Red Blood Cell (RBC) Count and Reticulocyte Count (RC)
Description: Blood samples were collected for the analysis of hematology parameters including RBC count and RC.
Time Frame: Days 1, 42 and 59
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 2 | 3
Trillion cells per liter
  RBC, Day 1, n=2, 3 | 3.45 (0.354) | 3.20 (0.300)
  RBC, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  RBC, Day 42, n=2, 2 | 3.30 (0.283) | 3.65 (0.071)
  RBC, Day 59, n=2, 3 | 3.35 (0.354) | 3.63 (0.493)
  RC, Day 1, n=2, 3 | 0.04090 (0.018102) | 0.06090 (0.038112)
  RC, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  RC, Day 42, n=2, 2 | 0.04610 (0.023052) | 0.07970 (0.057983)
  RC, Day 59, n=2, 3 | 0.03490 (0.014708) | 0.04580 (0.049537)

33. Other Pre Specified Outcome: Change From Baseline in Hematology Parameters of RBC Count and RC
Description: Blood samples were collected for the analysis of hematology parameters including RBC count and RC. Baseline value (Day 1) is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and at Days 42 and 59
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 2 | 3
Trillion cells per liter
  RBC, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  RBC, Day 42, n=2, 2 | -0.15 (0.071) | 0.60 (0.141)
  RBC, Day 59, n=2, 3 | -0.10 (0.000) | 0.43 (0.252)
  RC, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  RC, Day 42, n=2, 2 | 0.00520 (0.004950) | 0.00815 (0.010819)
  RC, Day 59, n=2, 3 | -0.00600 (0.003394) | -0.01510 (0.011467)

34. Other Pre Specified Outcome: Absolute Values of the Hematology Parameters of Hemoglobin and Mean Corpuscle Hemoglobin Concentration (MCHC)
Description: Blood samples were collected for the analysis of hematology parameters including hemoglobin and MCHC.
Time Frame: Days 1, 42 and 59
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Grams per deciliter
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 2 | 3
Grams per deciliter
  Hemoglobin, Day 1, n=2, 3 | 10.60 (0.849) | 9.77 (0.586)
  Hemoglobin, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Hemoglobin, Day 42, n=2, 2 | 10.45 (0.778) | 11.40 (0.424)
  Hemoglobin, Day 59, n=2, 3 | 10.40 (0.849) | 11.27 (1.002)
  MCHC, Day 1, n=2, 3 | 34.10 (0.000) | 34.23 (0.351)
  MCHC, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  MCHC, Day 42, n=2, 2 | 34.10 (0.141) | 33.75 (1.909)
  MCHC, Day 59, n=2, 3 | 34.00 (0.141) | 34.33 (1.447)

35. Other Pre Specified Outcome: Change From Baseline in Hematology Parameters- Hemoglobin and MCHC
Description: Blood samples were collected for the analysis of hematology parameters including hemoglobin and MCHC. Baseline value (Day 1) is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and at Days 42 and 59
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Grams per deciliter
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 2 | 3
Grams per deciliter
  Hemoglobin, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Hemoglobin, Day 42, n=2, 2 | -0.15 (0.071) | 1.85 (0.212)
  Hemoglobin, Day 59, n=2, 3 | -0.20 (0.000) | 1.50 (0.520)
  MCHC, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  MCHC, Day 42, n=2, 2 | 0.00 (0.141) | -0.65 (1.626)
  MCHC, Day 59, n=2, 3 | -0.10 (0.141) | 0.10 (1.127)

36. Other Pre Specified Outcome: Absolute Values of Hematology Parameter: Hematocrit
Description: Blood samples were collected for the analysis of hematology parameters including hematocrit.
Time Frame: Days 1, 42 and 59
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 2 | 3
Proportion of red blood cells in blood
  Day 1, n=2, 3 | 0.3105 (0.02616) | 0.2850 (0.01769)
  Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Day 42, n=2, 2 | 0.3065 (0.02475) | 0.3385 (0.00636)
  Day 59, n=2, 3 | 0.3065 (0.02475) | 0.3277 (0.03412)

37. Other Pre Specified Outcome: Change From Baseline in Hematology Parameter: Hematocrit
Description: Blood samples were collected for the analysis of hematology parameters including hematocrit. Baseline value (Day 1) is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and at Days 42 and 59
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 2 | 3
Proportion of red blood cells in blood
  Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Day 42, n=2, 2 | -0.0040 (0.00141) | 0.0615 (0.02192)
  Day 59, n=2, 3 | -0.0040 (0.00141) | 0.0427 (0.02212)

38. Other Pre Specified Outcome: Absolute Values of Hematology Parameter of Red Blood Cell Distribution Width (RDW)
Description: Blood samples were collected for the analysis of hematology parameters including RDW.
Time Frame: Days 1, 42 and 59
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Percentage of width
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 2 | 3
Percentage of width
  Day 1, n=2, 3 | 0.3105 (0.02616) | 0.2850 (0.01769)
  Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Day 42, n=2, 2 | 13.45 (0.212) | 14.00 (0.424)
  Day 59, n=2, 3 | 13.20 (0.141) | 13.70 (0.200)

39. Other Pre Specified Outcome: Change From Baseline in RDW
Description: Blood samples were collected for the analysis of hematology parameters including RDW. Baseline value (Day 1) is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and at Days 42 and 59
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Percentage of width
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 2 | 3
Percentage of width
  Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Day 42, n=2, 2 | 0.00 (0.424) | 1.15 (0.636)
  Day 59, n=2, 3 | -0.25 (0.354) | 0.70 (0.436)

40. Other Pre Specified Outcome: Absolute Values of the Hematology Parameter of Mean Corpuscular Hemoglobin (MCH)
Description: Blood samples were collected for the analysis of hematology parameters including MCH.
Time Frame: Days 1, 42 and 59
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 2 | 3
Picograms
  Day 1, n=2, 3 | 30.95 (0.354) | 30.67 (1.457)
  Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Day 42, n=2, 2 | 31.40 (0.424) | 31.40 (0.707)
  Day 59, n=2, 3 | 31.10 (0.141) | 30.93 (1.716)

41. Other Pre Specified Outcome: Change From Baseline in Hematology Parameter of MCH
Description: Blood samples were collected for the analysis of hematology parameters including MCH. Baseline value (Day 1) is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and at Days 42 and 59
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 2 | 3
Picograms
  Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Day 42, n=2, 2 | 0.45 (0.071) | -0.10 (0.990)
  Day 59, n=2, 3 | 0.15 (0.212) | 0.27 (0.862)

42. Other Pre Specified Outcome: Absolute Values of the Hematology Parameter of Mean Corpuscular Volume (MCV)
Description: Blood samples were collected for the analysis of hematology parameters including MCV.
Time Frame: Days 1, 42 and 59
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 2 | 3
Femtoliters
  Day 1, n=2, 3 | 91.0 (1.41) | 89.7 (3.51)
  Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Day 42, n=2, 2 | 92.0 (1.41) | 93.0 (2.83)
  Day 59, n=2, 3 | 91.5 (0.71) | 90.0 (3.00)

43. Other Pre Specified Outcome: Change From Baseline in Hematology Parameter of MCV
Description: Blood samples were collected for the analysis of hematology parameters including MCV. Baseline value (Day 1) is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and at Days 42 and 59
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 2 | 3
Femtoliters
  Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Day 42, n=2, 2 | 1.0 (0.00) | 1.5 (0.71)
  Day 59, n=2, 3 | 0.5 (0.71) | 0.3 (0.58)

44. Other Pre Specified Outcome: Absolute Values of Clinical Chemistry Parameters of Sodium, Potassium, Carbon-dioxide (Total), Chloride, Glucose and Urea
Description: Blood samples will be collected for the analysis of clinical chemistry parameters including; sodium, potassium, carbon-dioxide (total), chloride, glucose and urea.
Time Frame: Days 1, 42 and 59
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Millimoles per Liter
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 2 | 3
Millimoles per Liter
  Sodium, Day 1, n=2, 3 | 140.0 (1.41) | 136.7 (0.58)
  Sodium, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Sodium, Day 42, n=2, 2 | 139.5 (3.54) | 135.0 (7.07)
  Sodium, Day 59, n=2, 3 | 138.5 (0.71) | 136.0 (2.65)
  Potassium, Day 1, n=2, 3 | 4.70 (0.141) | 5.03 (0.757)
  Potassium, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Potassium, Day 42, n=2, 2 | 4.55 (0.495) | 5.15 (0.495)
  Potassium, Day 59, n=2, 3 | 4.45 (0.071) | 4.77 (0.306)
  Carbon-dioxide (total), Day 1, n=2, 3 | 20.5 (3.54) | 19.0 (3.46)
  Carbon-dioxide (total), Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Carbon-dioxide (total), Day 42, n=2, 2 | 22.0 (1.41) | 19.0 (0.00)
  Carbon-dioxide (total), Day 59, n=2, 3 | 22.5 (2.12) | 21.0 (2.00)
  Chloride, Day 1, n=2, 3 | 108.0 (0.00) | 105.7 (5.03)
  Chloride, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Chloride, Day 42, n=2, 2 | 108.0 (4.24) | 104.0 (9.90)
  Chloride, Day 59, n=2, 3 | 108.0 (2.83) | 104.7 (3.51)
  Glucose, Day 1, n=2, 3 | 7.60 (3.111) | 6.40 (4.424)
  Glucose, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Glucose, Day 42, n=2, 2 | 6.95 (2.333) | 12.50 (12.162)
  Glucose, Day 59, n=2, 3 | 7.45 (4.172) | 10.10 (7.066)
  Urea, Day 1, n=2, 3 | 18.00 (2.828) | 16.67 (5.508)
  Urea, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Urea, Day 42, n=2, 2 | 16.75 (2.475) | 21.00 (0.707)
  Urea, Day 59, n=2, 3 | 16.50 (0.707) | 19.33 (5.795)

45. Other Pre Specified Outcome: Change From Baseline in Clinical Chemistry Parameter: Sodium, Potassium, Carbon-dioxide (Total), Chloride, Glucose and Urea
Description: Blood samples will be collected for the analysis of clinical chemistry parameters including; sodium, potassium, carbon-dioxide (total), chloride, glucose and urea. Baseline value (Day 1) is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and at Days 42 and 59
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Millimoles per Liter
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 2 | 3
Millimoles per Liter
  Sodium, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Sodium, Day 42, n=2, 2 | -0.5 (4.95) | -1.5 (6.36)
  Sodium, Day 59, n=2, 3 | -1.5 (2.12) | -0.7 (2.31)
  Potassium, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Potassium, Day 42, n=2, 2 | -0.15 (0.354) | -0.05 (0.495)
  Potassium, Day 59, n=2, 3 | -0.25 (0.071) | -0.27 (0.503)
  Carbon-dioxide (total), Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Carbon-dioxide (total), Day 42, n=2, 2 | 1.5 (4.95) | 1.0 (4.24)
  Carbon-dioxide (total), Day 59, n=2, 3 | 2.0 (1.41) | 2.0 (2.00)
  Chloride, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Chloride, Day 42, n=2, 2 | 0.0 (4.24) | -2.0 (2.83)
  Chloride, Day 59, n=2, 3 | 0.0 (2.83) | 1.73 (1.73)
  Glucose, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Glucose, Day 42, n=2, 2 | -0.65 (0.778) | 4.25 (7.849)
  Glucose, Day 59, n=2, 3 | -0.15 (1.061) | 3.70 (3.477)
  Urea, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Urea, Day 42, n=2, 2 | -1.25 (5.303) | 3.00 (7.778)
  Urea, Day 59, n=2, 3 | -1.50 (3.536) | 2.67 (2.754)

46. Other Pre Specified Outcome: Absolute Values of Clinical Chemistry Parameters of Creatinine
Description: Blood samples will be collected for the analysis of clinical chemistry parameters including; creatinine.
Time Frame: Days 1, 42 and 59
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Micromoles per Liter
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 2 | 3
Micromoles per Liter
  Creatinine, Day 1, n=2, 3 | 246.65 (9.970) | 225.40 (74.164)
  Creatinine, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Creatinine, Day 42, n=2, 2 | 249.75 (15.627) | 272.25 (88.742)
  Creatinine, Day 59, n=2, 3 | 260.35 (8.132) | 245.17 (91.086)

47. Other Pre Specified Outcome: Change From Baseline in Clinical Chemistry Parameter: Creatinine
Description: Blood samples will be collected for the analysis of clinical chemistry parameters including; creatinine. Baseline value (Day 1) is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and at Days 42 and 59
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Micromoles per Liter
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 2 | 3
Micromoles per Liter
  Creatinine, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Creatinine, Day 42, n=2, 2 | 3.10 (5.657) | 36.70 (13.152)
  Creatinine, Day 59, n=2, 3 | 13.70 (18.102) | 19.77 (33.416)

48. Other Pre Specified Outcome: Absolute Values of Clinical Chemistry Parameters of Bilirubin (Direct/Indirect and Total)
Description: Blood samples will be collected for the analysis of clinical chemistry parameters including; bilirubin (direct/indirect and total).
Time Frame: Days 1, 14, 28, 42 and 59
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Micromoles per Liter
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 2 | 3
Micromoles per Liter
  Bilirubin total, Day 1, n=2, 3 | 5.0 (1.41) | 6.0 (0.00)
  Bilirubin total, Day 14, n=2, 3 | 5.0 (1.41) | 7.3 (1.15)
  Bilirubin total, Day 28, n=2, 3 | 6.0 (0.00) | 6.0 (0.00)
  Bilirubin total, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Bilirubin total, Day 42, n=2, 2 | 6.0 (0.00) | 9.0 (4.24)
  Bilirubin total, Day 59, n=2, 3 | 5.0 (1.41) | 6.7 (1.15)
  Direct Bilirubin, Day 1, n=2, 2: number analyzed (Participants) | 2 | 2
  Direct Bilirubin, Day 1, n=2, 2 | 1.0 (1.41) | 2.0 (0.00)
  Direct Bilirubin, Day 14, n=2, 2: number analyzed (Participants) | 2 | 2
  Direct Bilirubin, Day 14, n=2, 2 | 1.0 (1.41) | 2.0 (0.00)
  Direct Bilirubin, Day 28, n=2, 2: number analyzed (Participants) | 2 | 2
  Direct Bilirubin, Day 28, n=2, 2 | 1.0 (1.41) | 2.0 (0.00)
  Direct Bilirubin, Day 42, n=2, 1: number analyzed (Participants) | 2 | 1
  Direct Bilirubin, Day 42, n=2, 1 | 2.0 (0.00) | 2.0 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
  Direct Bilirubin, Day 59, n=2, 2: number analyzed (Participants) | 2 | 2
  Direct Bilirubin, Day 59, n=2, 2 | 2.0 (0.00) | 2.0 (0.00)
  Indirect Bilirubin, Day 1, n=2, 2: number analyzed (Participants) | 2 | 2
  Indirect Bilirubin, Day 1, n=2, 2 | 4.0 (0.00) | 4.0 (0.00)
  Indirect Bilirubin, Day 14, n=2, 2: number analyzed (Participants) | 2 | 2
  Indirect Bilirubin, Day 14, n=2, 2 | 4.0 (0.00) | 5.0 (1.41)
  Indirect Bilirubin, Day 28, n=2, 2: number analyzed (Participants) | 2 | 2
  Indirect Bilirubin, Day 28, n=2, 2 | 5.0 (1.41) | 4.0 (0.00)
  Indirect Bilirubin, Day 42, n=2, 1: number analyzed (Participants) | 2 | 1
  Indirect Bilirubin, Day 42, n=2, 1 | 4.0 (0.00) | 10.0 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
  Indirect Bilirubin, Day 59, n=2, 2: number analyzed (Participants) | 2 | 2
  Indirect Bilirubin, Day 59, n=2, 2 | 3.0 (1.41) | 5.0 (1.41)

49. Other Pre Specified Outcome: Change From Baseline in Clinical Chemistry Parameter: Bilirubin (Direct/Indirect and Total)
Description: Blood samples will be collected for the analysis of clinical chemistry parameters including; creatinine and bilirubin (direct/indirect and total). Baseline value (Day 1) is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and at Days 14, 28, 42 and 59
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Micromoles per Liter
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 2 | 3
Micromoles per Liter
  Bilirubin total, Day 14, n=2, 3 | 0.0 (0.00) | 1.3 (1.15)
  Bilirubin total, Day 28, n=2, 3 | 1.0 (1.41) | 0.0 (0.00)
  Bilirubin total, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Bilirubin total, Day 42, n=2, 2 | 1.0 (1.41) | 3.0 (4.24)
  Bilirubin total, Day 59, n=2, 3 | 0.0 (0.00) | 0.7 (1.15)
  Direct Bilirubin, Day 14, n=2, 2: number analyzed (Participants) | 2 | 2
  Direct Bilirubin, Day 14, n=2, 2 | 0.0 (0.00) | 0.0 (0.00)
  Direct Bilirubin, Day 28, n=2, 2: number analyzed (Participants) | 2 | 2
  Direct Bilirubin, Day 28, n=2, 2 | 0.0 (0.00) | 0.0 (0.00)
  Direct Bilirubin, Day 42, n=2, 1: number analyzed (Participants) | 2 | 1
  Direct Bilirubin, Day 42, n=2, 1 | 1.0 (1.41) | 0.0 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
  Direct Bilirubin, Day 59, n=2, 2: number analyzed (Participants) | 2 | 2
  Direct Bilirubin, Day 59, n=2, 2 | 1.0 (1.41) | 0.0 (0.00)
  Indirect Bilirubin, Day 14, n=2, 2: number analyzed (Participants) | 2 | 2
  Indirect Bilirubin, Day 14, n=2, 2 | 0.0 (0.00) | 1.0 (1.41)
  Indirect Bilirubin, Day 28, n=2, 2: number analyzed (Participants) | 2 | 2
  Indirect Bilirubin, Day 28, n=2, 2 | 1.0 (1.41) | 0.0 (0.00)
  Indirect Bilirubin, Day 42, n=2, 1: number analyzed (Participants) | 2 | 1
  Indirect Bilirubin, Day 42, n=2, 1 | 0.0 (0.00) | 6.0 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
  Indirect Bilirubin, Day 59, n=2, 2: number analyzed (Participants) | 2 | 2
  Indirect Bilirubin, Day 59, n=2, 2 | -1.0 (1.41) | 1.0 (1.41)

50. Other Pre Specified Outcome: Absolute Values of Clinical Chemistry Parameters of Alanine Transaminase (ALT), Alkaline Phosphatase (ALP) and Aspartate Transaminase (AST)
Description: Blood samples will be collected for the analysis of clinical chemistry parameters including; ALT, ALP and AST.
Time Frame: Days 1, 14, 28, 42 and 59
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: International units per Liter
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 2 | 3
International units per Liter
  ALT, Day 1, n=2, 3 | 21.0 (4.24) | 26.7 (7.02)
  ALT, Day 14, n=2, 3 | 15.0 (4.24) | 20.3 (6.81)
  ALT, Day 28, n=2, 3 | 15.5 (4.95) | 18.3 (8.08)
  ALT, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  ALT, Day 42, n=2, 2 | 16.0 (4.24) | 22.0 (9.90)
  ALT, Day 59, n=2, 3 | 20.5 (10.61) | 23.3 (8.08)
  ALP, Day 1, n=2, 3 | 113.5 (61.52) | 95.0 (42.44)
  ALP, Day 14, n=2, 3 | 97.0 (42.43) | 91.0 (33.87)
  ALP, Day 28, n=2, 3 | 99.5 (45.96) | 91.7 (38.40)
  ALP, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  ALP, Day 42, n=2, 2 | 99.0 (39.60) | 100.5 (37.48)
  ALP, Day 59, n=2, 3 | 108.5 (55.86) | 90.3 (29.26)
  AST, Day 1, n=2, 3 | 19.5 (7.78) | 21.7 (1.53)
  AST, Day 14, n=2, 3 | 16.5 (7.78) | 18.3 (3.51)
  AST, Day 28, n=2, 3 | 18.0 (9.90) | 18.7 (7.09)
  AST, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  AST, Day 42, n=2, 2 | 17.5 (10.61) | 16.5 (4.95)
  AST, Day 59, n=2, 3 | 20.5 (10.61) | 19.3 (6.03)

51. Other Pre Specified Outcome: Change From Baseline in Clinical Chemistry Parameter: ALT, ALP and AST
Description: Blood samples will be collected for the analysis of clinical chemistry parameters including; ALT, ALP and AST. Baseline value (Day 1) is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and at Days 14, 28, 42 and 59
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: International units per Liter
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 2 | 3
International units per Liter
  ALT, Day 14, n=2, 3 | -6.0 (0.00) | -6.3 (1.53)
  ALT, Day 28, n=2, 3 | -5.5 (0.71) | -8.3 (1.15)
  ALT, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  ALT, Day 42, n=2, 2 | -5.0 (0.00) | -5.0 (0.00)
  ALT, Day 59, n=2, 3 | -0.5 (6.36) | -3.3 (4.62)
  ALP, Day 14, n=2, 3 | -16.5 (19.09) | -4.0 (12.12)
  ALP, Day 28, n=2, 3 | -14.0 (15.56) | -3.3 (4.04)
  ALP, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  ALP, Day 42, n=2, 2 | -14.5 (21.92) | -6.5 (14.85)
  ALP, Day 59, n=2, 3 | -5.0 (5.66) | -4.7 (13.61)
  AST, Day 14, n=2, 3 | -3.0 (0.00) | -3.3 (2.08)
  AST, Day 28, n=2, 3 | -1.5 (2.12) | -3.0 (6.00)
  AST, Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  AST, Day 42, n=2, 2 | -2.0 (2.83) | -5.0 (2.83)
  AST, Day 59, n=2, 3 | 1.0 (2.83) | -2.3 (5.03)

52. Other Pre Specified Outcome: Absolute Values of Clinical Chemistry Parameters of Albumin
Description: Blood samples will be collected for the analysis of clinical chemistry parameters including; Albumin.
Time Frame: Days 1, 14, 28, 42 and 59
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Grams per Liter
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 2 | 3
Grams per Liter
  Day 1, n=2, 3 | 37.0 (5.66) | 41.7 (2.31)
  Day 14, n=2, 3 | 36.5 (2.12) | 40.7 (3.06)
  Day 28, n=2, 3 | 35.5 (3.54) | 39.3 (3.21)
  Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Day 42, n=2, 2 | 35.5 (3.54) | 38.5 (0.71)
  Day 59, n=2, 3 | 36.5 (6.36) | 40.3 (1.53)

53. Other Pre Specified Outcome: Change From Baseline in Clinical Chemistry Parameter: Albumin
Description: Blood samples will be collected for the analysis of clinical chemistry parameters including; Albumin. Baseline value (Day 1) is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and at Days 14, 28, 42 and 59
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Grams per Liter
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 2 | 3
Grams per Liter
  Day 14, n=2, 3 | -0.05 (0.354) | -0.10 (0.200)
  Day 28, n=2, 3 | -0.15 (0.212) | -0.23 (0.321)
  Day 42, n=2, 2: number analyzed (Participants) | 2 | 2
  Day 42, n=2, 2 | -0.15 (0.212) | -0.25 (0.354)
  Day 59, n=2, 3 | -0.05 (0.071) | -0.13 (0.153)

ADVERSE EVENTS:
Time Frame: Non-SAEs and SAEs were collected from the start of the treatment and Up to 59 days
Description: Non-SAEs and SAEs were collected in the Safety Population which comprised of participants who received at least one dose of study treatment.
Arm/Group | Daprodustat | Darbepoetin Alfa
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 0/2 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daprodustat (N=2) | Darbepoetin Alfa (N=3)
Faeces soft (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Bilateral foot discomfort secondary to Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Swollen right foot secondary to Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-08-07): https://cdn.clinicaltrials.gov/large-docs/12/NCT03446612/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-10): https://cdn.clinicaltrials.gov/large-docs/12/NCT03446612/SAP_001.pdf